CLINICAL TRIAL: NCT06120439
Title: Comparing the Quality of Recovery(QoR) of Pectoral Nerves(PECS) Block and General Anesthesia(GA) in Breast-conserving Surgery(BCS) With Sentinel Lymph Node Biopsy(SLNB):A Randomized Controlled Trial
Brief Title: Comparing the QoR of PECS Block and GA in Breast-conserving Surgery With Sentinel Lymph Node Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jun Zhang (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, Head of Department of Anesthesiology, Fudan University Shanghai Cancer Center, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSYDXSJLHLJSJ-1
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Pectoral Nerves Block; Breast-Conserving Surgery; Sentinel Lymph Node Biopsy
Keywords: Pectoral nerves block II; intercostal nerve block; dexmedetomidine; breast-conserving surgery; sentinel lymph node biopsy; quality of recovery
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, General; Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: The nerve block group was named the test group (T Group), and the laryngeal mask general anesthesia group was named the control group (C Group). The T Group received PECS II combined with intercostal nerve blockade, while the C Group underwent laryngeal mask insertion after general anesthesia induction.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The follow-up personnel and data analysts are blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T Group (Experimental): The T Group received PECS II(PMID: 22939099) combined with intercostal nerve block
  Interventions: Combination Product: PECS II combined with intercostal nerve blockade;
- C Group (Active Comparator): C Group underwent laryngeal mask insertion after general anesthesia induction.
  Interventions: Combination Product: General anesthesia with laryngeal mask

INTERVENTIONS:
Combination Product: PECS II combined with intercostal nerve blockade; — The patient was in a supine position, and under ultrasound guidance, the needle tip was first placed in the plane between the pectoralis major and minor muscles, and 10ml of 0.3% ropivacaine was injected. The needle was then advanced into the space between the pectoralis minor and serratus anterior muscles, and 20ml of 0.3% ropivacaine was injected. Intercostal nerve blockade: The range of intercostal blockade was determined based on the location of the breast surgery. The needle was inserted into the intercostal space from the posterior axillary line, and 3ml of 0.3% ropivacaine was injected into each intercostal space.
  Arms: T Group
Combination Product: General anesthesia with laryngeal mask — The C Group underwent general anesthesia induction using TCI propofol 3-3.5μg/ml, TCI remifentanil 1-2ng/ml, sufentanil 0.3μg/kg iv, midazolam 0.05mg/kg iv, and rocuronium 0.6mg/kg iv after loss of consciousness. After muscle relaxation, the laryngeal mask was inserted, and mechanical ventilation was performed with a tidal volume of 6ml/kg. Anesthesia maintenance included propofol 3-4μg/ml and remifentanil 1-2ng/ml.
  Arms: C Group

SUMMARY:
The aim of this randomized controlled trial (RCT) is to assess the Quality of Recovery (QoR) in Breast-conserving Surgery (BCS) with Sentinel Lymph Node Biopsy (SLNB) using Pectoral Nerves (PECS) Block and General Anesthesia (GA). The primary objectives are as follows: First, to determine if the PECS group exhibits better QoR; Second, to investigate if the PECS group experiences less postoperative pain and complications; Third, to examine if the PECS group demonstrates more stable hemodynamics.

DETAILED DESCRIPTION:
This study is a randomized controlled trial, with a 1:1 ratio for grouping. The experimental group is the T group, receiving Pecs II combined with intercostal nerve block, while the control group is the C group, receiving general anesthesia. The primary outcome measure is the QoR-15 score of the subjects 6 hours after surgery. Based on preliminary results, the control group had a QoR-15 score of 133±8 (n=6), and the experimental group needs to improve by at least 8 points (which is generally considered clinically significant, PMID:27159009). With a two-sided α=0.05 and a power of 99%, accounting for a 20% dropout rate, the final required sample size was calculated to be 96 cases, with 48 cases in each group.

If the proportion of dropout cases is less than 5% and considered "completely random missing," the missing records generated by the dropout cases will be directly excluded. Depending on the specific circumstances, either single imputation or multiple imputation methods will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for breast-conserving surgery with sentinel lymph node biopsy.
* Age between 18 and 70 years.
* Body Mass Index (BMI) < 30 kg/m2.
* American Society of Anesthesiologists (ASA) classification grade I-III.

Exclusion Criteria:

* Contraindications to regional anesthesia: site infection at the puncture site, allergy to local anesthetics, coagulation disorders, or bleeding risks.
* Impaired liver or kidney function.
* Pregnancy, lactation, possibility of pregnancy, or planned pregnancy.
* Preoperative use of analgesic drugs, history of chronic pain, or history of opioid abuse.
* Mental illness.
* Patients who refuse to participate.
* Patients deemed unsuitable for the clinical trial by the researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Postoperative QoR-15 at 6 hours | 6 hours after the surgery
  The 15-item quality of recovery(QoR-15) at 6 hours after the surgery.

SECONDARY OUTCOMES:
Postoperative NRS pain score at 6 hours | 6 hours after the surgery
  Postoperative numeric rating scales pain score at 6 hours after the surgery. Postoperative pain severity at rest and movement measured using a numerical rating scale(NRS) at 24 h. The numerical rating scale (NRS) is a line with numbers from 0 to 10 are spaced evenly across the page. And the NRS is bounded at the left-most end with "no pain" and at the right-most end with "worst pain imaginable". Pain levels below "4" are considered mild, "4-7" is moderate pain, and anything above "7" is considered severe pain. Patients are instructed to circle the number that represents the amount of pain that they are experiencing at the time of the evaluation. The movement status refers to maximum mobility of the upper arm of the surgical side. Remedial pain relief measures are initiated when the Numeric Rating Scale (NRS) score exceeds 4.
The number of patients who experience intraoperative hypotension | From the beginning of anesthesia to the end of the surgery.
  During the surgery and anesthesia process, MAP ≤ 65 mmHg is defined as intraoperative hypotension. Record the number of patients who experience intraoperative hypotension.
Changes in hemodynamics (mean arterial pressure) after the surgical incision. | From the beginning of anesthesia to three minutes after the surgical incision.
  Monitor the magnitude of hemodynamic changes compared to baseline after the incision. The main comparison is the magnitude of changes in mean arterial pressure between the two groups.
Changes in hemodynamics (heart rate) after the surgical incision. | From the beginning of anesthesia to three minutes after the surgical incision.
  Monitor the magnitude of hemodynamic changes compared to baseline after the incision. The main comparison is the magnitude of changes in heart rate between the two groups.

OTHER OUTCOMES:
Postoperative QoR-15 at 2 hours | 2 hours after the surgery
  The 15-item quality of recovery(QoR-15) at 2 hours after the surgery.
Postoperative QoR-15 at 24 hours | 24 hours after the surgery
  The 15-item quality of recovery(QoR-15) at 24 hours after the surgery.
Postoperative NRS pain score at 2 hours | 2 hours after the surgery
  Postoperative numeric rating scales pain score at 2 hours after the surgery. Postoperative pain severity at rest and movement measured using a numerical rating scale(NRS) at 24 h. The numerical rating scale (NRS) is a line with numbers from 0 to 10 are spaced evenly across the page. And the NRS is bounded at the left-most end with "no pain" and at the right-most end with "worst pain imaginable". Pain levels below "4" are considered mild, "4-7" is moderate pain, and anything above "7" is considered severe pain. Patients are instructed to circle the number that represents the amount of pain that they are experiencing at the time of the evaluation. The movement status refers to maximum mobility of the upper arm of the surgical side. Remedial pain relief measures are initiated when the Numeric Rating Scale (NRS) score exceeds 4.
Postoperative NRS pain score at 24 hours | 24 hours after the surgery
  Postoperative numeric rating scales pain score at 24 hours after the surgery. Postoperative pain severity at rest and movement measured using a numerical rating scale(NRS) at 24 h. The numerical rating scale (NRS) is a line with numbers from 0 to 10 are spaced evenly across the page. And the NRS is bounded at the left-most end with "no pain" and at the right-most end with "worst pain imaginable". Pain levels below "4" are considered mild, "4-7" is moderate pain, and anything above "7" is considered severe pain. Patients are instructed to circle the number that represents the amount of pain that they are experiencing at the time of the evaluation. The movement status refers to maximum mobility of the upper arm of the surgical side. Remedial pain relief measures are initiated when the Numeric Rating Scale (NRS) score exceeds 4.
The number of patients requiring additional analgesics | 24 hours after the surgery
  The number of patients requiring additional analgesics for rescue analgesia after the surgery is completed.
the number of patients who experience post-operative hypotension. | 24 hours after the surgery
  MAP ≤ 65 mmHg is defined as hypotension. Record the number of patients who experience intraoperative hypotension.
the number of patients who experience intraoperative Bradycardia. | From the beginning of anesthesia to the end of the surgery.
  During the surgery and anesthesia process, a heart rate below 45 bpm is defined as intraoperative Bradycardia. Record the number of patients who experience intraoperative Bradycardia.
the number of patients who experience post-operative Bradycardia. | 24 hours after the surgery
  A heart rate below 45 bpm is defined as Bradycardia. Record the number of patients who experience Bradycardia.
Proportion of patients experiencing postoperative nausea and vomiting | 24 hours after the surgery
  Proportion of patients experiencing postoperative nausea and vomiting at least once at 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No